CLINICAL TRIAL: NCT02821117
Title: An Evaluation of Self-Management of Diabetes Using FreeStyle Libre Flash Glucose Monitoring System in Young People
Brief Title: FreeStyle Libre Glucose Monitoring System Paediatric Study
Acronym: SELFY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADC-UK-PMS-16028
Record Dates: First submitted 2016-06-27; First posted 2016-07-01 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus, Paediatric; Sensing Technology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): FreeStyle Libre Flash Glucose Monitoring System
  Interventions: Device: FreeStyle Libre Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Subjects will wear the FreeStyle Libre Flash Glucose Monitoring System masked for 14 days followed by 8 weeks unmasked wear.
  During the 2 weeks of masked device wear participants will use the BG strip port for self-monitoring of blood glucose (SMBG). Scanning the sensor at least every 8 hours during this phase.
  Followed by 8 weeks of unmasked device wear when participants will use the device (Sensor glucose and SMBG) according to labelling for their day to day management.

SUMMARY:
The study is designed to determine glycaemic control achieved using the FreeStyle Libre Flash Glucose Monitoring System (FreeStyle Libre) versus Self-Monitoring Blood Glucose (SMBG) for the self-management of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥4 years and ≤17 years.
* Has an identified Caregiver of ≥18 years.
* Type 1 diabetes using insulin (administered by injections or CSII) for at least 1 year.
* Current insulin regimen has been unchanged for at least 2 months prior to enrolment (e.g. change of insulin or administration method), with no plans to change insulin regimen.
* Currently testing BG, on average at least 2 times per day.

Exclusion Criteria:

* Concomitant disease or condition that may compromise patient safety including and not limited to; cystic fibrosis, severe mental illness, known or suspected eating disorder or any uncontrolled long term medical condition.
* Currently prescribed oral steroid therapy for any acute or chronic condition (or requires it during the study).
* Currently receiving dialysis treatment or planning to receive dialysis during the study.
* Female participant known to be pregnant.
* Participating in another device or drug study that could affect glucose measurements or glucose management.
* Currently using or planning to use FreeStyle Libre Flash Glucose Monitoring System or a Continuous Glucose Monitoring (CGM) device during the study.
* Has used the FreeStyle Libre Flash Glucose Monitoring System or a Continuous Glucose Monitoring (CGM) device in the previous 3 months.
* Known (or suspected) allergy to medical grade adhesives.
* In the investigator's opinion the participant is unsuitable to participate due to any other cause/reason (participant and caregiver considered).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Time in Range | Baseline and days 56 to 70
  Time in range (Sensor glucose 3.9-10.0 mmol/L [70-180 mg/dL]) in days 56-70 minus time in range at baseline (days 1-15).

CONTACTS AND LOCATIONS:
Locations (10):
- Kinder- und Jugendkrankenhaus, Hanover, Germany
- Ireland (2):
  - National Children's Hospital, Dublin
  - Temple Street Children's University Hospital, Dublin
- United Kingdom (7):
  - Royal Belfast Hospital for Sick Children, Belfast, County Antrim
  - Antrim Area Hospital, Antrim
  - Ulster Hospital, Belfast
  - St. James University Hospital, Leeds Teaching Hospitals NHS Trust, Leeds
  - Altnagelvin Hospital, Londonderry
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Southampton University Hospital NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided